CLINICAL TRIAL: NCT06483412
Title: Evaluation Tobacco Prevention Toolkit Healthy Futures: Alternative-to-Suspension Vaping Intervention
Brief Title: An Evaluation of the Tobacco Prevention Toolkit Healthy Futures: Alternative-to-Suspension Vaping Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: California School-Based Health Alliance (Other)
Responsible Party: Principal Investigator, Bonnie Halpern-Felsher, Marron and Mary Elizabeth Kendrick Professor in Pediatrics II, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-75499
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Use Cessation; Addiction
Keywords: Tobacco Use; Tobacco Use Cessation; E-Cigarette Use; Suspension
MeSH Terms: conditions — Tobacco Use Cessation; Behavior, Addictive; Tobacco Use; Vaping

STUDY DESIGN:
Intervention Model Description: Employs a step-wedged design that involves delay-of-treatment for the control group. Prognostic blocks of schools will be assigned to treatment (10 schools) versus delay-in-treatment (10 schools) in Year 1 of the intervention. In Years 2 and 3, the 10 schools that served as "control" schools will cross over and implement the Healthy Futures: Alternative-to-Suspension intervention.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stanford REACH Lab Healthy Futures Curriculum (Experimental): At the start of Year 1, schools will be randomized in a 1:1 ratio to either receive 'Stanford REACH Lab's Healthy Futures: Alternative-to-Suspension Curriculum' or 'delay-in-treatment (standard of care)'. Students in these schools who are found using tobacco/nicotine or who want to quit these products will be administered the Healthy Futures: Alternative-to-Suspension curriculum for 3 years.
  Interventions: Behavioral: Healthy Futures: Alternative-to-Suspension Curriculum
- Delay In Treatment (Experimental): At the start of Year 1, schools will be randomized in a 1:1 ratio to either receive 'Stanford REACH Lab's Healthy Futures: Alternative-to-Suspension Curriculum' or 'delay-in-treatment (standard of care).' Schools in this arm will receive a standard of care for one year. After year 1, the delay-in-treatment group will crossover to receive 'Stanford REACH Lab's Healthy Futures: Alternative-to-Suspension Curriculum until year 3 (receive intervention for years 2 and 3).
  Interventions: Behavioral: Healthy Futures: Alternative-to-Suspension Curriculum

INTERVENTIONS:
Behavioral: Healthy Futures: Alternative-to-Suspension Curriculum — Healthy Futures: Alternative-to-Suspension Curriculum uses a trauma-informed and restorative practice lens and uses principles of motivational interviewing (MI) and cognitive-behavioral therapy (CBT) to help students understand the harms of nicotine, reduce stress, increase positive coping, and provide resources to quit.

SUMMARY:
The Healthy Futures: Alternative-to-Suspension Curriculum is a free, online curriculum developed to educate students and provide them with resources to quit tobacco/nicotine use. The investigation aims to estimate the extent to which Healthy Futures: Alternative-to-Suspension changes high school student's knowledge of, attitudes towards, intentions to use, and actual use of tobacco/nicotine.

DETAILED DESCRIPTION:
Youth who use tobacco/nicotine products on school campuses are often detained, suspended, or expelled. Healthy Futures: Alternative-to-Suspension is an online curriculum that uses principles of motivational interviewing and cognitive behavioral therapy, incorporating a restorative practice and trauma-informed lens.

The goals of the study are three-fold: (1) Assess changes in the perspectives of school administrators, educators, counselors, and health staff around the feasibility, acceptability, and usefulness of implementing Healthy Futures: Alternative-to-Suspension as an appropriate and effective response to tobacco use on campus (including versus suspension or expulsion); (2) Assess high school students' acceptability and perceptions of Healthy Futures: Alternative-to-Suspension; and (3) Estimate the extent to which Healthy Futures: Alternative-to-Suspension changes high school students' knowledge of, attitudes towards, intentions/susceptibility to use, and actual use of tobacco/nicotine products. The Stanford REACH Lab and California School-Based Health Alliance (CSHA) will partner to evaluate Healthy Futures: Alternative-to-Suspension using a school-based randomized waitlist-controlled trial in 20 high schools in California (n = 10 Healthy Futures: Alternative-to-Suspension treatment schools and 10 control schools).

ELIGIBILITY:
Inclusion criteria for schools

* Agree to be randomized to use the Healthy Futures: Alternative-to-Suspension curriculum or to use their current standard of care exclusive of Healthy Futures: Alternative-to-Suspension
* Agree that teachers, counselors, or other school personnel will schedule an online survey prior to and after implementation of Healthy Futures: Alternative-to-Suspension or current standard of care with students caught using e-cigarettes or other tobacco products and with students self-reporting use of those products and seeking help to quit
* Has access to a school nurse/school health officer/school counselor or school psychologist
* Agree that parental consent, where required, will be sought from students prior to survey administration.
* Agree that the study is in the wider interest of the public health of adolescents and in their schools interest.

Inclusion criteria for participants Adolescents, aged 14-18, from grades 9-12, who are agreeable to participate in the study and provide assent.

Exclusion Criteria:

Adolescents, aged 14-18 years, from grades 9-12 who do not speak English.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2540 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in tobacco/nicotine use | Baseline, follow-up 1 (following intervention at one year), follow-up 2 (6 months post-intervention), follow-up 3 (6 months past follow-up 2), and follow-up 4 (6 months past follow-up 3) up to 2.5 years of the study.
  Investigator-originated survey measures (questions) ever tobacco/nicotine use and past 30-day tobacco/nicotine use. All students in both arms will be asked to complete a survey at baseline (just before treatment), follow-up 1 (immediately post-intervention), follow-up 2 (6 months after completing intervention), and so on every 6 months for 2.5 years of the study.

SECONDARY OUTCOMES:
Change in intention of tobacco/nicotine use scale score | Baseline, follow-up 1 (following intervention at one year), follow-up 2 (6 months post intervention), follow-up 3 (6 months past follow-up 2), and follow-up 4 (6 months past follow-up 3) up to 2.5 years of the study.
  Participants will self-report changes in their intention/susceptibility to use tobacco/nicotine products using a validated four-point scale in a survey. This survey measures changes in intention to use tobacco/nicotine with questions related to the participant's knowledge of and resistance to the use of tobacco/nicotine products.
  Susceptibility is measured by the following questions:
  1. Have you ever been curious about using an e-cigarette?
  2. Do you think that you will try an e-cigarette soon?
  3. If one of your best friends were to offer you an e-cigarette, would you use it?"
  Response options for all three questions included a four-point scale: "Definitely yes," "Probably yes," "Probably not," and "Definitely not."

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Halpern-Felsher, Ph.D, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No